CLINICAL TRIAL: NCT02253927
Title: Phase I Sequential Dose Escalation Study of Pharmacokinetics, Safety and Tolerability After Single Dose (225 Mg-450 mg) Oral Administration of BILR 355 (SDS) Plus Low-dose Ritonavir in Healthy Volunteers
Brief Title: Dose Escalation Study of Pharmacokinetics, Safety and Tolerability After Single Dose Administration of BILR 355 (SDS) Plus Low-dose Ritonavir in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1188.32
Record Dates: First submitted 2014-09-30; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — Ritonavir

ARMS (1):
- BILR 355 (dose escalation) + Ritonavir (Experimental): escalating dose groups, for food effect evaluation lowest dose group (D1) with high fat meal breakfast after wash-out period
  Interventions: Drug: BILR 355 - D1; Drug: BILR 355 - D2; Drug: BILR 355 - D3; Drug: BILR 355 - D4; Drug: Ritonavir; Other: high fat breakfast

INTERVENTIONS:
Drug: BILR 355 - D1
Drug: BILR 355 - D2
Drug: BILR 355 - D3
Drug: BILR 355 - D4
Drug: Ritonavir
Other: high fat breakfast

SUMMARY:
The primary objective was to explore the relative bioavailability of increasing doses of BILR 355 BS, as a sodium dodecyl sulfate-containing solid formulation (SDS), in combination with ritonavir 100 mg and to explore the dose-concentration proportionality of increasing doses.

A secondary objective was to explore the effect of food on the pharmacokinetics of BILR 355 (SDS)

ELIGIBILITY:
Inclusion Criteria:

1. Males or females who met the inclusion/exclusion criteria, females who are not pregnant nor nursing, and who agreed to use a double-barrier method of birth control (condoms or diaphragm plus spermicide) throughout the trial (alone or in addition to other methods of birth control such as oral contraceptives)
2. Healthy HIV negative adult volunteers
3. Age ≥18 and ≤60 years
4. BMI ≥18.5 and BMI ≤29.9 kg/m2
5. Ability to give signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local regulations

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Surgery of gastrointestinal tract (except appendectomy)
3. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
4. History of relevant orthostatic hypotension, fainting spells or blackouts
5. Chronic or relevant acute infections
6. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
7. Intake of drugs with a long half-life (>24 hours) within at least one month prior to study drug administration and during the trial
8. Use of drugs within 10 days prior to administration or during the trial which might reasonably influence the results of the trial
9. Participation in another trial with an investigational drug within two months prior to administration or during the trial
10. Current smoker
11. Alcohol abuse (more than 60 g/day)
12. Drug abuse (positive urine test for illicit prescription or non-prescription drugs or drugs of abuse)
13. Blood donation (more than 100 mL within four weeks prior to study drug administration or during the trial)
14. Excessive physical activities (within one week prior to study drug administration or during the trial)
15. Any laboratory value outside the reference range that is of clinical relevance at screening, according to the judgment of the investigator
16. Inability to comply with dietary regimen required by the protocol
17. Infected with hepatitis B or hepatitis C viruses (defined as either being hepatitis B surface antigen, or hepatitis C antibody positive)
18. Pregnant or lactating females

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2006-05; Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
AUC0-inf (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 120 hours after drug administration
Cmax (Maximum measured concentration of the analyte in plasma) | up to 120 hours after drug administration
AUC0-tz (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | up to 120 hours after drug administration
CL/F (Apparent clearance of the analyte in plasma following extravascular administration) | up to 120 hours after drug administration
Tmax (Time from dosing to the maximum concentration of the analyte in plasma) | up to 120 hours after drug administration
t½ (Terminal half-life of the analyte in plasma) | up to 120 hours after drug administration

SECONDARY OUTCOMES:
Number of patients with adverse events | up to 10 days after last dose administration